CLINICAL TRIAL: NCT06497829
Title: Geranylgeraniol Supplementation in Patients With Mevalonate Kinase Deficiency, MVK Deficiency (hyperIgD Syndrome)
Brief Title: Geranylgeraniol Supplementation in Patients With Mevalonate Kinase Deficiency
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Motol (Other)
Collaborators: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Anna Sediva, Prof. Anna Sediva, MD, PhD, University Hospital, Motol
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: EK-30/22
Record Dates: First submitted 2024-07-01; First posted 2024-07-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Mevalonate Kinase Deficiency
Keywords: immunoglobulin D; mevalonate kinase; isoprenoids; geranylgeraniol
MeSH Terms: conditions — Mevalonate Kinase Deficiency | interventions — geranylgeraniol

STUDY DESIGN:
Intervention Model Description: Patients with MVK deficiency compared to healthy controls and to subjects on statin therapy (statins target the same metabolic pathway)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients with MVK deficiency (Experimental): patients fulfilling inclusion criteria
  Interventions: Dietary Supplement: geranylgeraniol

INTERVENTIONS:
Dietary Supplement: geranylgeraniol — GG Pure (Extendlife Natural Products) containing GG gold®30 Annatto Extract, 500 mg capsule, use for 3 months, once daily

SUMMARY:
Mevalonate kinase deficiency (HyperIgD syndrome, HIDS) is an inborn error of immunity caused by a block in the mevalonate pathway. The subsequent lack of isoprenoids with antiinflammatory properties might contribute to the autoinflammatory nature of the disease.

A pilot study aims to verify the safety and efficacy of the dietary supplement Geranylgeraniol, aiming at a mitigation of isoprenoids deficiency caused by the above-mentioned block in the MVK pathway.

DETAILED DESCRIPTION:
Mevalonate kinase (MVK) deficiency, a rare autosomal recessive disease, significantly impacts metabolism and immunity, leading to mevalonic aciduria in severe cases and hyper-IgD syndrome (HIDS) in partial deficiency. These conditions arise due to disruptions in the mevalonate pathway, which is an essential metabolic pathway responsible for the synthesis of non-sterol isoprenoids and other molecules. The resulting metabolic blockade triggers autoinflammatory responses, primarily due to deficient isoprenoid intermediates such as geranylgeranyl pyrophosphate (GGPP).

This study evaluates the safety and efficacy of dietary geranylgeraniol (GG) supplementation in patients with genetically confirmed mevalonate kinase deficiency.

The pilot study consists of a month of a pre-supplementation period to monitor the level of inflammation and clinical status in patients with MVK deficiency(HIDS).

This period is followed by 3 months of supplementation of 150mg of GeranylGraniol (GG Pure (Extendlife Natural Products) containing GG gold®30 Annatto Extract, 500 mg capsule (30% geranylgeraniol, 150 mg per capsule).

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 12 years with genetically confirmed MVK deficiency
* Overall good clinical status apart from the clinical presentation of the MVK deficiency
* Normal liver tests
* Compliance with the study protocol

Exclusion Criteria:

• Children below 12 years

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2022-01-25 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in inflammatory parameters | 3 monhts of intervention
  Monitoring inflammatory markers before and after intervention - CRP (C reactive protein) and SAA (serum amyloid A) levels will be measured before and after the intervention (time 0 and time 3 months of GG use).
  These values tend to be elevated in patients with MVK deficiency due to their inflammatory status compared to normal values defined in clinical laboratories (UHMotol CRP < 8 mg/l, SAA < 10 mg/l).
  The expected outcome would result in a decrease in inflammatory markers.

SECONDARY OUTCOMES:
Change in the clinical status of patients | 3 months
  Monitoring of general clinical status and defined parameters - general condition, fatigue, fever, skin manifestations, abdominal pain, and headache using a questionnaire. The questionnaire is designed for daily monitoring of the parameters mentioned above. The scale of the questionnaire is from 1 to 10, with 1 being the best, normal condition, and 10 being the worst degree of disability.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Šedivá, Mgr, Principal Investigator — University Hospital, Motol
Locations (1):
- University Hospital, Motol, Prague, Czechia

IPD SHARING:
Plan to Share IPD: Undecided
anonymized patient data consisting of clinical and laboratory sets of follow-up parameters are shared with participating researchers